CLINICAL TRIAL: NCT02207894
Title: A Survey on the Success of Inhibitor Elimination Using Individualized Concentrate Selection and Controlled (High Dose) Immune Tolerance Induction (ITI)
Brief Title: A Survey on the Success of Inhibitor Elimination Using Individualized Concentrate Selection and Controlled ITI
Status: Recruiting | Type: Observational
Sponsor: Haemophilia Centre Rhine Main (Other)
Collaborators: University of Bonn (Other); Skane University Hospital (Other); Hopital Cardiologique Louis Pradel, Unité d'Hemostase Clinique Bron (Unknown)
Responsible Party: Sponsor
Other Study IDs: HZRM_ObsITI_4th Am.Version
Record Dates: First submitted 2014-05-06; First posted 2014-08-04 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Haemophilia A
Keywords: Haemophilia A, factor VIII, development of inhibitor
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, plasma.
Oversight: Data Monitoring Committee: No

SUMMARY:
This research program is initiated to evaluate and document data on the success of ITI in 300 haemophilia A patients with newly developed or already existing FVIII-inhibitors (also patients who might potentially have failed in earlier ITIs), which will be treated with ITI - preferably high-dose based on individualized product selection, in order to improve management of this potentially devastating complication of haemophilia treatment.

In order to investigate the role of in vitro tests on individual ITI success rate in patients undergoing ITI, the inhibitor plasma samples can be assayed against different FVIII concentrates using the following in vitro tests: Batch selection, Thrombin generation assay (TGA), Thrombin Generation Test (TGT) to monitor FVIII efficacy, Epitope mapping,IgG Subclasses specific for FVIII, Immunogenotyping.

DETAILED DESCRIPTION:
As a result of many technological advances in the last two decades, current factor VIII (FVIII) concentrates (both plasma-derived and recombinant products) are considered very safe in terms of pathogen safety.

The development of inhibitors against FVIII or factor IX (FIX) is considered as a major complication during replacement therapy of haemophiliacs.

Prospective studies of previously untreated patients (PUPs) have suggested that inhibitors develop in up to 33% of patients with moderate to severe haemophilia A. Several strategies are used to control bleedings in such patients, e.g. high-dose treatment with FVIII concentrates, treatment with activated prothrombin complex concentrate (aPCC) or treatment with activated factor VII (FVIIa).

Immune tolerance induction (ITI) in order to eradicate inhibitors in patients suffering from an inhibitor to FVIII with high dose treatment of FVIII was first reported in 1977 by Brackmann & Gormsen in the so-called "Bonn Protocol" and was investigated from then on in a series of clinical studies applying the same or a modified version of the "Bonn Protocol". During these investigations high dose FVIII treatment has been proven efficacious in inducing immune tolerance and was shown to exert a long lasting effect in more than 80 % of the patients treated.

The observational immune tolerance induction research program (ObsITI) will allow a systematic prospective and retrospective data documentation and analysis on the success rate of ITI by using individualized concentrate selection.

Pre-ITI-phase:

Aim of this evaluation is to assess current pre-ITI treatment strategies in inhibitor patients from detection of inhibitor until start of ITI (early start vs. delayed start) and the effect of pre-ITI treatment (prophylaxis and on-demand treatment in case of bleeds/surgery) with bypassing agents (rFVIIa, NovoSeven®, aPCC, FEIBA®, emicizumab, Hemlibra®) and / or FVIII on the titre at start of ITI, on the success rate of ITI, the number of break-through bleeds and life-threatening bleeds.

ObsITI-Rescue ITI Study:

Patients who fail FVIII-stand-alone ITI or who are no candidates for FVIII-stand-alone ITI and who are treated with ITI regimens including immunosuppressive agents can be included in this sub-study. Aim of this study is to document ITI regimens including immunosuppressive therapy (Rituximab, steroids, mycophenolate mofetil/MMF, sirolimus or other immunosuppressive agents) combined with regular FVIII administration, potential drug related side effects, outcome and duration of immune tolerance (relapse and recurrence of inhibitors).

Optional sub-studies:

In order to investigate the role of in vitro tests on individual ITI success rate in patients undergoing ITI, the inhibitor plasma samples can be assayed against different FVIII concentrates using the following in vitro tests:

1. Batch selection: The potential variation in inhibitor reactivity with different FVIII concentrates/batches of the same concentrate can optionally be studied according to a modified Oxford method (HZRM Hämophilie-Zentrum Rhein Main, Germany).
2. Thrombin generation assay (TGA): In this optional in vitro test the plasma samples from an inhibitor patient can be spiked with different concentrates and the thrombin generation will be measured using the TGA to evaluate the potential of different FVIII concentrates to generate thrombin (Haemophilia Centre Malmö, Sweden).
3. Thrombin Generation Test (TGT): TGT will evaluate the correlation between clinical bleeding phenotype of patients and their thrombin generation capacity before ITI in order to predict the patients with the highest risk of bleeding. In vitro efficacy of two FVIII doses (low and high) in the presence and absence of FEIBA® and emicizumab will be evaluated (Louis Pradel Cardiology Hospital, Bron, France).
4. Epitope mapping / IgG Subclasses: The isotypic antibody epitopes on FVIII will be identified in plasma samples from inhibitor patients. This will help to identify relevant epitopes recognised by inhibitors in haemophilia A. This research program will give an opportunity to comprehensively study various aspects of inhibitors and the induction of immunetolerance in a relevant number of patients. Knowledge about relevant epitopes from patient plasma rather than from model systems (i.e. monoclonal antibodies or mouse models) will help to understand the immune response to FVIII and to develop novel strategies to deplete inhibitors or inhibitor secreting B cells (Haemophilia Centre, University Hospital Bonn, Germany). Plasma samples will also be tested for IgG-subclasses specific for FVIII. Most inhibitors belong to the subclasses IgG1 and IgG4. There are some indications that the ratio of IgG1 and IgG4 might influence ITI outcome (Haemophilia Centre, University Hospital Bonn, Germany).
5. Immunogenotyping / HLA Genotyping: In addition, this study will investigate genetic risk factors (gene defect responsible for haemophilia, HLA class II alleles, immune response genes) as a potential variable with impact on course and outcome of ITI. Recently a significantly higher inhibitor incidence has been found in patients (brothers) with IL-10.G allele 134, TNFα - 308G>A polymorphism within Hap and polymorphisms in the CTLA-4-gene compared to those brothers without the above mentioned polymorphisms (Haemophilia Centre, University Hospital Bonn, Germany).

If patients do not respond to FVIII stand-alone ITI and any immune modulating/ immunosuppressive agents are added to ITI,ITI courses can be followed up in the ObsITI-Rescue ITI sub-study. Immunosuppressive therapy has to be documented as concomitant medication. Follow up visits should be done in the same intervals as with stand-alone FVIII-ITI.

ELIGIBILITY:
Inclusion Criteria:

* Based on the decision of the treating physicians in the participating centres, male patients at any age suffering from severe (FVIII activity < 1%), moderate (FVIII activity >1% - 5%), or mild (FVIII activity > 5%) haemophilia A will be included into this post marketing observation if relevant inhibitor levels (> 0.6 BU) have been detected, or - in case of an inhibitor level <0.6 BU - with reduced recovery or half-life of FVIII.
* The observation is also open for patients who failed an earlier ITI attempt.

Exclusion Criteria:

* Female

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all male patients with haemophilia A and inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-08; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of ITI, the primary endpoint of this observation, is defined according to the following criteria (The measure is a composite).: Inhibitor titre <0.6 BU, Incremental recovery of FVIII in the normal range,Half-life of FVIII > 7 hours. | one year
  The efficacy of ITI, the primary endpoint of this observation, is defined according to the following criteria (The measure is a composite):
  * Inhibitor titre <0.6 BU (at least 2 consecutive determinations)
  * Incremental recovery of FVIII in the normal range (> 80% of normal) with samples taken prior to and 15 or 30 minutes after FVIII treatment.
  * Half-life of FVIII > 7 hours (blood samples for FVIII determination should be taken prior to and 15 or 30 minutes, 1, 2, 4, 8 and either 12 or 24 hours after FVIII treatment.
  Complete Success:
  All three criteria above met.
  Partial Success:
  Two of the three criteria above met.
  Partial Response:
  One of the three criteria above met.
  Partial Failure of ITI-treatment:
  Inhibitor still present, but titre has decreased to <5 BU.
  Complete Failure of ITI-treatment:
  None of the above mentioned criteria met, and the inhibitor titre is still ≥5 BU.

SECONDARY OUTCOMES:
The following secondary endpoints will also be evaluated.The measure is a composite. | one year
  The following secondary endpoints will be evaluated:
  * the success rates of the different types of products selected for ITI, especially those of pure and VWF-stabilized FVIII concentrates
  * the maintenance in case of complete or partial ITI success
  * the clinical relevance of the individual in vitro testing and batch selection, the selected type of concentrate will be correlated with the ITI success
  * the adverse drug reactions and possibly ITI efficacy related events occurring during the ITI-treatment phase
  * the compliance with the ITI-treatment regimen
  * the time necessary to achieve complete or partial success of individualized ITI
  * the impact of inhibitor titres at start of ITI and during the course of ITI, including the peak titre of the inhibitor
  * the number of break-through bleeding events during the course of ITI-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escuriola Ettingshausen, MD, Principal Investigator — Director HZRM
Locations (1):
- Haemophilia Centre Rhine Main, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Click here for more information about this study:The Observational Immune Tolerance Induction (ObsITI) research program — http://www.obsiti.de